CLINICAL TRIAL: NCT01625728
Title: A Comparison of Vocal Demands With Vocal Performance Among Classroom Teachers
Brief Title: Vocal Demands Among Classroom Teachers
Status: Completed | Type: Observational
Sponsor: Southern Illinois University Carbondale (Other)
Responsible Party: Sponsor
Other Study IDs: 10529
Record Dates: First submitted 2012-03-14; First posted 2012-06-21 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2018-08

CONDITIONS: Voice Disorders
Keywords: Voice; aerodynamics; acoustics
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental group.: Participants are either student teachers or practicing teachers.
- Control Group.: Participants are no students teachers or practicing teachers.

SUMMARY:
The purpose of the study "A comparison of vocal demands with vocal performance among classroom teachers" is to gather information about the voice production of teachers using three separate strategies: (a) measures of voice assessed with the Computerized Speech Lab (CSL) and the Phonatory Aerodynamic System (PAS) instruments in the SIUC Voice Lab.

DETAILED DESCRIPTION:
(a) measures of voice assessed with the Computerized Speech Lab (CSL) and the Phonatory Aerodynamic System (PAS) instruments in the SIUC Voice Lab

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in teaching education programs; active teachers.

Exclusion Criteria:

* Current diagnosed with voice disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the experimental group: student teachers enrolled in teaching education programs and active teachers. Participants in the control group: not enrolled in teaching education programs and are not active teachers.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Acoustic measures of voice. | 1 year
  Acoustic measures of voice (i.e., fundamental frequency, total phonation time, and SPL. Participants will be tested three separate times distributed in equal periods throughout one academic semester (i.e., 16 weeks).

SECONDARY OUTCOMES:
Identify changes in aerodynamic measures of voice. | 1 year
  Identify changes in aerodynamic measures of voice (airflow). Participants will be tested three separate times distributed in equal periods throughout one academic semester (i.e., 16 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Claudia Franca, Ph.D., Principal Investigator — Southern Illinois University Carbondale
Locations (1):
- Southern Illinois University Carbondale, Carbondale, Illinois, United States

IPD SHARING:
Plan to Share IPD: No